CLINICAL TRIAL: NCT06770738
Title: Predictive Performance of EuroSCORE-II and POSPOM for Perioperative Mortality in Cardiac Surgery: A Retrospective Study
Brief Title: EuroSCORE-II and POSPOM in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kerem Erkalp, MD, Prof, professor, Istanbul University - Cerrahpasa
Other Study IDs: 017
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Disease; Cardiovascular Diseases; Cardiovascular Complication; Anesthesia; Perioperative/Postoperative Complications; Surgery
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operation group: Patients aged 18 and over, patients who have CABG surgery, valve surgery or both, and patients with on-pump surgery in 2020-2024 will be included in the study. The sample size was calculated as 314 with an effect size of 0.2, 95% power and 0.05 error level using the G Power 3.1.9.2 package program, taking into account the study of Kaplan et al.
  Interventions: Other: There is no intervention in this study.

INTERVENTIONS:
Other: There is no intervention in this study. — This study is planned as a retrospective study. Only the information of the patients will be used.

SUMMARY:
We aim to compare the performances of the European System for Cardiac Operative Risk Evaluation (EuroSCORE-II) and the PreOperative Score to Predict Postoperative Mortality (POSPOM) in predicting in-hospital mortality among patients undergoing on-pump cardiac surgery, with further evaluation of discrimination, calibration, agreement, and clinical utility.

This retrospective observational study will be conducted at a single tertiary university cardiac surgery centre. Adult patients (≥18 years) who underwent coronary artery bypass grafting, valve surgery, or combined procedures between 2020 and 2024 will be included. No experimental interventions will be applied. Preoperative EuroSCORE-II and POSPOM values will be calculated for all patients. Discrimination will be assessed using ROC and precision-recall curves with DeLong's test. Calibration will be evaluated using calibration-in-the-large, calibration slope, Hosmer-Lemeshow testing, and GiViTI calibration belts. Agreement will be analyzed using ICC, CCC, Bland-Altman plots, and Passing-Bablok and Deming regression. Subgroup analyses will be performed by age and sex.

DETAILED DESCRIPTION:
Preoperative risk assessment is important in determining the treatment plans of patients who will undergo surgery, providing patient education for the postoperative period, providing insight into prognosis, and determining healthcare quality standards. The European System for Cardiac Operative Risk Evaluation-II (EuroSCORE-II) was developed specifically for patients in cardiac surgery. It is a scoring system widely used worldwide that predicts mortality through preoperative evaluation. New studies in the literature have reported that the sensitivity of EuroSCORE-II may be lower in older patients (over 70 and 80 years of age). A scoring system with higher predictive power is aimed by making modifications to EuroSCORE-II or by making comparisons with other scoring systems. PreOperative Score to Predict Post-Operative Mortality (POSPOM), defined by Le Manach et al. in 2016, is a useful scoring system that can be used for all types of surgery and can predict postoperative mortality through preoperative evaluation of patients. POSPOM includes parameters that evaluate the patient's age, the type of surgery to be performed, and the patient's comorbidities. It appears to be a useful scoring system because it is applicable to all types of surgery and provides information about patient mortality in a short time by collecting patient values in 3 main groups. There are various studies conducted on patients undergoing hip fractures, radical cystectomy, uro-oncological surgery, and non-cardiac vascular surgery. However, a review of the literature revealed an absence of studies investigating cardiac surgery patients alone.

The primary objective of this study was to investigate whether the POSPOM score has sufficient predictive power for in-hospital mortality in patients undergoing cardiac surgery. The secondary objective was to evaluate the correlation between POSPOM mortality predictions and EuroSCORE-II mortality predictions in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over, patients who have CABG surgery, valve surgery or both, and patients with on-pump surgery will be included in the study.

Exclusion Criteria:

* . Patients under the age of 18, patients with off-pump surgery, and patients with non-cardiac vascular surgery will be excluded from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Turkish people including all genders at the age of 18-99 and was operated open heart surgery will be the study population.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
investigation whether the POSPOM score has sufficient predictive power for in-hospital mortality in patients undergoing cardiac surgery | 1 month
  The primary objective of this study was to investigate whether the POSPOM score has sufficient predictive power for in-hospital mortality in patients undergoing cardiac surgery.
  Measure Type: Continuous Unit of Measure: ROC-AUC
  Minimum: 0.50 Maximum: 1.00
  Description of Meaningful Outcome:
  Predictive performance will be considered clinically meaningful if the ROC-AUC of the POSPOM score for in-hospital mortality is significantly greater than 0.50.

SECONDARY OUTCOMES:
Correlation of EuroSCORE-II and POSPOM | 15 days
  Evaluation of the correlation between POSPOM mortality predictions and EuroSCORE-II mortality predictions in patients undergoing cardiac surgery.
  Measure Type: Continuous Unit of Measure: Correlation coefficient (r)
  Minimum: -1.0 Maximum: +1.0
  Description of Meaningful Outcome:
  A statistically significant correlation coefficient (p < 0.05) will indicate agreement between POSPOM and EuroSCORE-II mortality predictions. A correlation coefficient of |r| ≥ 0.50 will be considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Erkalp, Dr, Principal Investigator — Professor
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)